CLINICAL TRIAL: NCT04881279
Title: Maintaining Optimal Trauma Outcomes: Resilience in the Midst of a Ransomware Attack
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Weidun Alan Guo, MD, PhD, Department of Surgery, State University of New York at Buffalo
Other Study IDs: STUDY00002779
Record Dates: First submitted 2021-04-21; First posted 2021-05-11 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2021-05

CONDITIONS: Trauma; Electronic Health Record
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Trauma admissions in April-June 2016.
- Ransomware Group: Trauma admissions in April-June 2017.
  Interventions: Other: Event

INTERVENTIONS:
Other: Event — Ransomware attack
  Groups: Ransomware Group

SUMMARY:
Retrospective review of de-identified hospital emergency room and trauma registry data and operating room case logs from April 9th through June 9th, 2016, 2017 examining outcomes as affected by a ransomware attack in a level I trauma center

DETAILED DESCRIPTION:
On April 9, 2017, Erie County Medical Center, Western New York's sole level I trauma center was under cyberattack. The perpetrators utilized ransomware that gained access to the hospital's web server and encrypted hospital data, forcing a system-wide downtime for nearly 2 months. Electronic medical records, imaging, and interdepartmental communication were severely affected, forcing the hospital to temporarily return to pre-EMR era operations. We examined the impact of this cyber disaster on the outcomes of trauma care.

Retrospective review of de-identified hospital emergency room and trauma registry data and operating room case logs from April 9th through June 9th, 2016, 2017, and 2018. Baseline characteristics of study cohort for each period will be examined using the chi-square test for categorical variables and the Student's t-test for continuous variables that are normally distributed.

This was an exempt study in our institution.

ELIGIBILITY:
Inclusion Criteria:

* All trauma patient admissions that were seen through the ECMC Trauma Center from April to June 2016 and April to June 2017
* Adult patients >13 years old

Exclusion Criteria:

-Patients who came through the emergency department that were not categorized as trauma patients

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Trauma patients being served by the level I trauma center catchment area in Western New York, Southern Ontario (Canada), and Northern Pennsylvania
Sampling Method: Non-Probability Sample
Enrollment: 846 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Hospital and ICU length of stay (LOS), and in-hospital mortality | April to June 2016 and 2017
  Hospital and ICU length of stay (LOS) in days And in-hospital mortality between cohorts expressed as percentage of cohort

SECONDARY OUTCOMES:
Disposition at discharge and AHRQ patient safety indicators: DVT/PE, CLABSI, CAUTI, and organ/space surgical infection. | April to June 2016 and 2017
  Disposition at discharge defined as either discharged home, died, or sent to a rehabilitation facility, all expressed as the proportion of the cohort group with the above-mentioned findings reported in percentages
  All AHRQ patient safety indicators: DVT/PE, CLABSI, CAUTI, and organ/space surgical infection are indicated as the proportion of the cohort group with the above-mentioned findings reported in percentages

CONTACTS AND LOCATIONS:
Overall Officials: W. Alan Guo, MD, PhD, Principal Investigator — State University of Buffalo
Locations (1):
- Erie County Medical Center, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No